CLINICAL TRIAL: NCT06835179
Title: Evaluation of the Efficacy and Safety of SBRT Combined With CAPEOX, Bevacizumab, and PD-1 Inhibitor in RAS-Mutant, MSS-Type, and Unresectable Metastatic Colorectal Cancer: a Single-center, Single-arm, Open-label Clinical Trail.
Brief Title: SBRT Combined With CAPEOX, Bevacizumab, and PD-1 Inhibitor for the Treatment of RAS-Mutant, MSS-Type, Unresectable Metastatic Colorectal Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRSYM202502
Record Dates: First submitted 2025-02-11; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Unresectable Metastatic Colorectal Cancer; Microsatellite Stable (MSS) Colorectal Cancer (CRC); RAS-mutant Colorectal Cancer
Keywords: SBRT; CAPEOX; Bevacizumab; PD-1 Inhibitor; RAS-Mutant; Microsatellite Stable (MSS); Unresectable Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Spinocerebellar Degenerations; Colorectal Neoplasms | interventions — Immune Checkpoint Inhibitors; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients first receive short-course SBRT (total dose of 30-60 Gy, completed in 3-5 fractions). Within two weeks after SBRT, the liver function and other toxicity reactions of patients are closely monitored to ensure they can tolerate subsequent drug treatment. Then, patients proceed to drug therapy: each treatment cycle lasts for 21 days, including intravenous administration of tislelizumab (200mg on day 1), bevacizumab (7.5mg/kg on day 1), oxaliplatin (135mg/m² on day 1), as well as oral capecitabine (1g/m² twice daily from day 1 to day 14). Up to six cycles of induction therapy may be administered
  Interventions: Radiation: SBRT; Drug: PD-1 Inhibitors; Drug: CapeOX + bevacizumab

INTERVENTIONS:
Radiation: SBRT — SBRT short course radiotherapy (total dose 30-60 Gy, completed in 3-5 sessions)
Drug: PD-1 Inhibitors — Tislelizumab (200mg on day 1)
Drug: CapeOX + bevacizumab — intravenous administration of bevacizumab (7.5mg/kg on day 1), oxaliplatin (135mg/m² on day 1), as well as oral capecitabine (1g/m² twice daily from day 1 to day 14)

SUMMARY:
SBRT Combined with CAPEOX, Bevacizumab, and PD-1 Inhibitor in RAS-Mutant, Microsatellite Stable (MSS), Unresectable Metastatic Colorectal Cancer (mCRC): a Single-center, Single-arm, Open-label Clinical Trail

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is currently one of the most common malignant tumors of the digestive tract in clinical practice. According to the latest cancer data in China, CRC ranks as the fourth leading cause of cancer-related deaths, with both its incidence and mortality rates showing an increasing trend. The early diagnosis and treatment rates of CRC in China remain significantly lower compared to developed countries. Most patients are diagnosed at locally advanced or metastatic stages, resulting in poor treatment outcomes and prognosis. Among newly diagnosed cases, 20% already present with distant metastases (metastatic colorectal cancer, mCRC), with a 5-year survival rate below 20%.

The NCCN and CSCO guidelines recommend standard treatments for mCRC patients, including fluorouracil-, oxaliplatin-, and/or irinotecan-based chemotherapy regimens combined with angiogenesis-targeting agents (e.g., bevacizumab) or epidermal growth factor receptor (EGFR)-targeted therapies (e.g., cetuximab), depending on the patient's RAS and BRAF status. RAS mutations are present in 50-56% of mCRC cases. For RAS-mutant mCRC patients, bevacizumab combined with chemotherapy is the standard first-line treatment. However, these patients exhibit poorer prognoses and shorter survival times compared to those with RAS wild-type mCRC. Studies also indicate that RAS-mutant mCRC features an immunosuppressive tumor microenvironment. Thus, enhancing the efficacy of first-line therapy for this subgroup remains a major clinical challenge.

In recent years, immune checkpoint inhibitors (ICIs) have revolutionized treatment paradigms for several solid cancers, including melanoma and lung cancer, by inducing durable responses and significantly improving outcomes. Microsatellite instability-high (MSI-H) CRC, characterized by high tumor mutational burden and neoantigen production, activates the immune system and demonstrates high responsiveness to ICIs. Multiple immunotherapies have been approved for MSI-H CRC, markedly prolonging survival and improving quality of life. However, microsatellite stable (MSS) mCRC, accounting for approximately 95% of cases, is considered an immunologically "cold tumor" due to low tumor mutational burden and limited immune cell infiltration. Only a small subset of MSS patients, such as those with POLE/POLD1 mutations, may benefit from ICIs, whereas monotherapy with ICIs shows minimal efficacy in most MSS/pMMR tumors. Consequently, novel strategies are urgently needed to enhance immunotherapy responses in this subgroup.

Radiotherapy not only improves local tumor control by directly killing irradiated tumor cells but also activates systemic antitumor immunity through multiple mechanisms, potentially reducing metastatic risk and synergizing with immunotherapy. First, radiotherapy promotes the release of pro-phagocytic signals (e.g., calreticulin) while downregulating anti-phagocytic signals like CD47, enhancing macrophage-mediated tumor phagocytosis. Post-radiotherapy release of high-mobility group box 1 (HMGB1) and upregulation of MHC-I expression facilitate tumor antigen processing and presentation to CD8+ T cells. Additionally, radiation-induced DNA damage may generate neoantigens and trigger immune surveillance. Studies show that DNA repair-deficient tumor cells exhibit growth suppression in immunocompetent mice post-radiotherapy, a phenomenon absent in immunodeficient models, suggesting that accumulated mutations in repair-deficient cells increase neoantigen burden and drive immune responses. Radiation may also elevate mutational load, providing novel targets for immune recognition. Furthermore, radiotherapy modifies the tumor stromal microenvironment by inducing cytokine production. For instance, radiation promotes TNF release, significantly reducing myeloid-derived suppressor cell (MDSC) infiltration, while enhancing CXCL9/CXCL10 secretion to recruit cytotoxic T cells. Collectively, these mechanisms shift the immune milieu toward tumor elimination, providing a rationale for combining radiotherapy with immunotherapy.

Against this backdrop, we designed this study: Evaluation of the Efficacy and Safety of SBRT Combined with CAPEOX, Bevacizumab, and PD-1 Inhibitor in RAS-Mutant, Microsatellite Stable (MSS), and Unresectable Metastatic Colorectal Cancer (mCRC) : a Single-center, Single-arm, Open-label Clinical Trail.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, regardless of gender.
* Lower edge of the lesion located ≥12 cm from the anal verge.
* Histologically confirmed colorectal adenocarcinoma.
* Confirmed as unresectable by multidisciplinary team (MDT) evaluation.
* RAS mutation-positive.
* Microsatellite/mismatch repair status: MSS/pMMR.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival ≥3 months.
* Adequate hematological, hepatic, and renal function:

Neutrophil count ≥1.5 × 10⁹/L; Platelet count ≥75 × 10⁹/L; Serum total bilirubin ≤1.5 × upper normal limit (UNL); Aspartate aminotransferase (AST) ≤2.5 × UNL; Alanine aminotransferase (ALT) ≤2.5 × UNL; Serum creatinine ≤1.5 × UNL.

* Karnofsky Performance Status (KPS) score ≥70.
* Adequate organ function with no contraindications to surgery, radiotherapy, chemotherapy, or immunotherapy.
* No prior chemotherapy or other antitumor therapy before enrollment.
* No prior immunotherapy received.
* Willingness and ability to comply with the study protocol during the trial period.
* Signed written informed consent.

Exclusion Criteria:

* Patients who have received antibodies against programmed death receptor-1 (PD-1) or its ligand (PD-L1), as well as antibodies against cytotoxic T lymphocyte associated antigen 4 (CTLA-4).
* Patients with any active autoimmune diseases or a history of requiring steroid or immunotherapy treatment.
* Complex situations with concurrent active bleeding, perforation, or requiring emergency surgery.
* Have received systemic anti-cancer treatment for rectal cancer.
* Simultaneously present with other non colorectal cancer tumor diseases.
* Patients with interstitial lung disease, non infectious pneumonia or uncontrollable systemic diseases (such as diabetes, hypertension, pulmonary fibrosis and acute pneumonia).
* Any grade 2 or above toxic reactions (classified according to the Common Terminology Criteria for Adverse Events (CTCAE) 5th edition) caused by previous treatment that have not subsided (excluding anemia, hair loss, and skin pigmentation).
* Pregnant or lactating women.
* Patients who are known or have been tested for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
* Known or suspected history of allergies to any relevant drugs used in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR rate) | 1 year
  ORR is defined as the proportion of patients who achieve the best objective response, either complete response (CR) or partial response (PR), according to the RECIST criteria (version 1.1).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 1 year
  DCR is defined as the proportion of patients who achieve complete response (CR), partial response (PR), or disease stability (SD) according to the RECIST criteria (version 1.1).
Progression Free Survival (PFS) | 2 years
  PFS is defined as the time from enrollment to the first recording of disease progression, or the time of death from any cause, whichever occurs earlier.

IPD SHARING:
Plan to Share IPD: No